CLINICAL TRIAL: NCT06804681
Title: Is Intraoperative PTH Monitoring Obsolete in Times of Choline PET/CT?
Brief Title: Is Intraoperative PTH Monitoring Obsolete in Times of Choline PET/CT? a Prospective Multicenter Cohort Study to Determine Whether the Regular Preoperative Use of Choline-PET/CT Scan Obviate the Need for Intraoperative PTH-measurement in Patients with Primary Hyperparathyreoidism
Status: Not yet recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01785
Record Dates: First submitted 2025-01-03; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Histology Blood values
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
In patients with primary hyperparathyreoidism (pHPT) in 80-90% only one of the four parathyroid glands has developed an autonomy and is causative for the disease. Localisation diagnostics are used to help identify the affected gland or glands in order to enable more focused surgical approaches and reduce morbidity of the surgery, as well as operative time. The gold standard for imaging in Germany and Austria are sonography and scintigraphy. If imaging is not conclusive, Choline-PET/CT, which has been shown to have a higher specificity than the scintigraphy, especially for multiglandular disease, is performed mostly in Austria, but only on special indications in Germany. In Switzerland, as of 2023 the Choline-PET/CT has replaced the scintigraphy and is routinely performed in patients with indication for parathyroidectomy in many hospitals.

The current S2k guideline recommends to perform an intraoperative PTH measurement before and 10 minutes after removal of the parathyroid gland in order to assess the success of the surgery. Due to the short half-life of PTH of around three minutes, a PTH drop of 50% or into the normal range within 10 minutes of removal of the suspected gland has a high sensitivity and specificity for cure. If PTH drop is inadequate, further gland exploration is performed. The intraoperative measurement of PTH is associated with waiting time in the OR and uncertainty if the next patient can be anesthetized, prolonging surgeries by 30-60 minutes depending on the local facilities. If the Choline-PET/CT is sufficiently sensitive and specific in detecting both uni- and multiglandular disease, surgery according to Choline-PET/CT findings could make waiting for intraoperative PTH drop unnecessary.

The aim of the study is to determine whether the regular use of Choline-PET/CT can obviate the need for intraoperative PTH-measurement with the potential to shorten the length of parathyroid surgeries. This could save considerable costs and justify the regular use of Choline-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* pHPT, preoperative Choline-PET, intraoperative PTH

Exclusion Criteria:

* no consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pHPT
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Determine the successful removal of all parathyroid glands responsible for the pHPT based on the preoperative Choline-PET/CT findings with measurement of parathormone and calcium level | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland